CLINICAL TRIAL: NCT05233826
Title: Phase 1 Study Evaluating the Safety and Immunogenicity of COVI-VAC as a Booster Dose in Previously Vaccinated Adults Against COVID-19
Brief Title: Safety and Immunogenicity of COVI-VAC as a Booster Dose in Adults Previously Vaccinated Against COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codagenix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDX-CoV-002
Record Dates: First submitted 2022-02-03; First posted 2022-02-10 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: Covid-19 vaccines; Covid-19 vaccine booster shot; Heterologous prime boost; COVID-19 vaccination; Vaccines, attenuated
MeSH Terms: conditions — COVID-19 | interventions — COVI-VAC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COVI-VAC (Experimental): COVI-VAC Nose Drops
  Interventions: Biological: COVI-VAC

INTERVENTIONS:
Biological: COVI-VAC — Intranasal, live attenuated vaccine against SARS-CoV-2

SUMMARY:
The purpose of this study is to to evaluate the safety and immune response of COVI-VAC given as a single booster dose in healthy adults previously vaccinated against COVID-19 with an authorised mRNA or adenovirus-vectored vaccine. Approximately 30 participants who have been fully vaccinated ≥ 3 months ago will be enrolled and receive one dose of COVI-VAC. COVI-VAC is administered by drops into each nostril. To assess the safety of the vaccine, each participant will record symptoms and oral temperature in a diary daily for 7 days after receiving COVI-VAC or placebo.

During the full study safety laboratory tests, physical exams, and vital signs (including oxygen saturation) will be conducted periodically for safety. Adverse events and medication use will be recorded.

Blood samples and intranasal samples will be collected periodically to assess the immune response from the vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 65 years of age, inclusive, on the day of signing the ICF
2. Body mass index (BMI) ≤ 35 kg/m2
3. In good health with no history, or current evidence, of clinically significant medical conditions with particular reference to, but not restricted to, thromboembolic disorders, coronary heart disease, chronic obstructive lung disease, and no clinically significant test abnormalities that will interfere with participant safety, as defined by medical history, physical examination, vital signs (including oxygen saturation), and safety laboratory tests as determined by the Investigator
4. Previous receipt of an authorised mRNA or adenovirus-vectored COVID-19 vaccine with completion of vaccine regimen ≥ 3 months before Day 1

Exclusion Criteria:

1. Residents of residential care facilities
2. Pregnant or lactating women
3. Inadequate venous access for repeated phlebotomy
4. History of confirmed or suspected SARS-CoV-2 infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Humoral Immunogenicity | Day 1
  IgG Titer measured by ELISA on day 1
Humoral Immunogenicity | Day 1
  IgG Titer measured by ELISA on day 29
Humoral Immunogenicity | Day 181
  IgG Titer measured by ELISA on day 181
Humoral Immunogenicity measured by neutralizing antibodies | Day 1
  neutralising antibody titer measured by microneutralisation assay in serum on days 1
Humoral Immunogenicity measured by neutralizing antibodies | Day 29
  neutralising antibody titer measured by microneutralisation assay in serum on day 29
Humoral Immunogenicity measured by neutralizing antibodies | Day 181
  neutralising antibody titer measured by microneutralisation assay in serum on day 181

SECONDARY OUTCOMES:
Vaccine and Virus Shedding | Day 4
  SARS-CoV-2 genome copy number/mL as assessed by quantitative polymerase chain reaction (qPCR) assay in nasopharyngeal swab samples collected on Day 4
Vaccine and Virus Shedding | Day 8
  SARS-CoV-2 genome copy number/mL as assessed by quantitative polymerase chain reaction (qPCR) assay in nasopharyngeal swab samples collected on Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- HMR, London, United Kingdom